CLINICAL TRIAL: NCT06463171
Title: Phase II Clinical Study of Almonertinib in Combination With Lastet in the First-line Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer With EGFR Mutations
Brief Title: Phase II Trial of Almonertinib Plus Lastet for EGFR+ Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of the Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024LY0323
Record Dates: First submitted 2024-06-10; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer Non-small Cell Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy (Experimental): Almonertinib, dosing regimen: 110mg/day orally, once daily in a 28-day cycle, continuously.
  Lastet, dosing regimen: 50 mg/day orally, every 28 days in a cycle, two weeks of continuous oral administration, two weeks off.
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib, dosing regimen: 110mg/day orally, once daily in a 28-day cycle, continuously.
  Lastet, dosing regimen: 50 mg/day orally, every 28 days in a cycle, two weeks of continuous oral administration, two weeks off.
  Other Names: Lastet

SUMMARY:
The goal of this clinical trial is to test in Locally Advanced or Metastatic Non-small Cell Lung Cancer patients with EGFR Mutations. The main question it aims to answer is:

Evaluation of the Efficacy and Safety of Aumolertinib in Combination with Lastet for the Treatment of EGFR-Mutated Locally Advanced or Metastatic Non-small Cell Lung Cancer in First-line Therapy.

Participants will be treated with a combination of Aumolertinib and Lastet.

ELIGIBILITY:
Inclusion Criteria:

* Prior to the implementation of any trial-related procedures, written informed consent must be obtained.
* Age ≥18 years.
* Patients with locally advanced (Stage III B/III C), metastatic, or recurrent (Stage IV) non-small cell lung cancer (NSCLC) confirmed histologically or cytologically, who are ineligible for surgical intervention and cannot undergo curative radiochemotherapy, as per the 8th edition TNM staging classification of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer.
* Provide archived tumor tissue or tissue obtained from biopsy at screening for biomarker testing, including EGFR mutation status, etc.;
* Presence of EGFR positive mutation;
* Investigator confirmation of at least one measurable lesion according to RECIST 1.1 criteria.
* Patients who have previously received platinum-containing adjuvant chemotherapy/radiotherapy, neoadjuvant chemotherapy/radiotherapy, or radical radiochemotherapy for advanced disease, with disease progression occurring >6 months after the last treatment, may participate in this study;
* Expected life expectancy ≥3 months.
* ECOG PS 0-1.
* Adequate hematologic function, defined as an absolute neutrophil count ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90g/L (without a history of blood transfusion in the past 7 days).
* Adequate liver function, defined as total bilirubin level ≤1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 times ULN for all patients, or for patients with liver metastasis, AST and ALT levels ≤5 times ULN.
* Adequate renal function, defined as serum creatinine ≤1.5 times ULN.
* Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; if a subject is on anticoagulant therapy, INR/PT should be within the therapeutic range set by the anticoagulant.
* Women of childbearing potential must undergo a pregnancy test within 7 days prior to the start of treatment, with negative results; and reliable contraception methods (such as intrauterine devices, oral contraceptives, and condoms) should be used during the trial and for 30 days after the end of the trial. Men of childbearing potential should use condoms for contraception during the trial and for 30 days after the end of the trial.
* Willingness to comply with regular follow-up visits and adhere to trial requirements.

Exclusion Criteria:

* 1. Currently participating in an interventional clinical study treatment;
* Have previously received anti-EGFR treatment;
* Received traditional Chinese medicine with antitumor indications or immunomodulatory drugs (such as thymosin, interferon, interleukin, etc.) within 2 weeks before the first dose;
* Have a history of allergic reactions to any of the study drug components.
* Have active hemoptysis (more than half a teaspoon), active diverticulitis, abdominal abscess, gastrointestinal obstruction, and peritoneal metastasis;
* Have tumor compression of surrounding vital organs (such as the esophagus) with accompanying related symptoms, compression of the superior vena cava, or invasion of major mediastinal vessels, the heart, etc.;
* Known to have brain metastases. Patients judged by the investigator to be asymptomatic or have stable brain metastases may be enrolled;
* Have active systemic infections, including tuberculosis (clinical diagnosis including medical history, physical examination, imaging findings, and TB testing according to local medical routines), hepatitis B (known to be HBV surface antigen (HBsAg) positive, with HBV DNA ≥1000cps/ml or the lower limit of the reference value), hepatitis C, or human immunodeficiency virus (HIV antibody positive);
* Known to have mental illness or substance abuse that may affect compliance with trial requirements;
* Recently treated with a full dose of oral or non-oral anticoagulants or thrombolytics. Prophylactic use of anticoagulants is allowed.
* Have a medical history, disease, treatment, or laboratory abnormality that may interfere with the trial results or prevent the subject from participating in the study throughout, or the investigator considers participation in the study not to be in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | up to 24 months
  PFS is defined as the period from the start of treatment until the disease progresses or the patient dies from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Disease Control Rate | 24 months
  Disease Control Rate (DCR) is to describe the proportion of patients who have achieved a response to treatment that includes not only complete and partial responses but also stable disease.
Duration of Response | 24 months
  The Duration of Response (DoR) is a clinical measure to determine the length of time that a tumor continues to respond to treatment without the cancer worsening.
Objective Response Rate | 24 months
  The Objective Response Rate (ORR) is a key metric used in oncology to assess the proportion of patients in a study or treatment group who achieve an objective response (CR or PR).
Overall Survival | up to 24 months
  OS is measured from the date of the initiation of treatment to the date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chunxia Su, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - Zhongshan hospital, Shanghai
  - The First Affiliated Hospital of Xiamen University, Xiamen

IPD SHARING:
Plan to Share IPD: No
In clinical trials, it is essential to strictly protect the privacy of patients' personal information. Data sharing may inappropriately increase the risk of privacy breaches, especially when data anonymization is not handled properly. Additionally, researchers or sponsors, based on their considerations of data ownership and intellectual property rights, have the authority to decide whether and how to share the data.

REFERENCES:
- [Derived] Chen J, Wang L, Liu L, Zhao J, Wu Y, Yu X, Su C. Aumolertinib in combination with Lastet in the first-line treatment of EGFR-mutated, locally advanced or metastatic non-small cell lung cancer (EVOLUTION): protocol for a single-arm, phase II clinical trial. BMJ Open. 2025 Apr 29;15(4):e097576. doi: 10.1136/bmjopen-2024-097576. PMID 40306921